CLINICAL TRIAL: NCT00743951
Title: Feasibility Study: Does Screening Plus Patient Decision Aids Reduce Unnecessary Surgical Referrals for Total Joint Arthroplasty in Practices With Long Waiting Lists for Surgical Consults?
Brief Title: Feasibility Study: Effect of Patient Decision Aids for Total Joint Replacement on Surgical Referrals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other); University of Ottawa (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OHREB 2006724-01H
Record Dates: First submitted 2007-07-25; First posted 2008-08-29 (Estimated); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis
Keywords: patient decision aids; patient preferences; osteoarthritis; joint replacement; waiting times
MeSH Terms: conditions — Osteoarthritis; Patient Preference

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Patient decision aid (Experimental): Patient decision aid about treatment options for osteoarthritis
  Interventions: Behavioral: 1 Patient decision aid; Behavioral: 2 Usual care
- 2 Usual care (Active Comparator): Usual patient educational materials
  Interventions: Behavioral: 2 Usual care

INTERVENTIONS:
Behavioral: 1 Patient decision aid — Patients will receive:
  i)patient education booklet ii) a video/DVD PtDA for either hip (Treatment choices for hip osteoarthritis) or knee (Treatment choices for knee osteoarthritis) © Health Dialog 2005.
  iii) a personal decision form is an interactive form used by patients after the DVD to elicit their knowledge, values, preferred option, and perceptions of the decision making process.
  iv) Referral to the surgeon with a standardized report of their clinical findings plus decisional data (knowledge, values, preference).
  Arms: 1 Patient decision aid
Behavioral: 2 Usual care — Patient will be given i) education booklet from local hospital which is a standardized teaching booklet given to all patients describing preparation for surgery, recovery after surgery, discharge plans.
  ii) Referral to the surgeon with a standardized report of their clinical findings.

SUMMARY:
Ministries of Health consider wait lists for total joint replacement a top priority. Research priorities to manage wait lists indicate the need to establish benchmarks that consider patient preferences. However, patients' preferences for hip or knee replacements are strongly associated with their misperceptions of the indicators for, and the risks and benefits of, these procedures. These misperceptions can be corrected with the use of patient decision aids. When decision aids are used in combination with assessing surgical eligibility, there may be a reduction in unnecessary referrals for surgery either because the patient is ineligible or because the eligible candidates make informed decisions to forgo this option.

The study objective is to pilot test the feasibility of a trial evaluating the effects of patient decision aids on reducing unnecessary surgical referrals for total joint replacement, when used in combination with a general practitioner run clinic to screen patients with hip or knee osteoarthritis for surgical eligibility.

The investigators expect to provide evidence of feasibility (e.g. ease of recruiting patients, delivering the interventions, measuring patient outcomes) and sample size needed for a larger scale study. This study should also provide evidence for planning implementation of the interventions and standardized training across other centers.

DETAILED DESCRIPTION:
Background:

Current research priorities to manage wait times for total joint arthroplasty (TJA) indicate the need to establish benchmarks that consider patient preferences. Among clinically appropriate candidates for this procedure, patients' preferences for surgery is very low; between 8.5 and 14.9% of clinically ideal candidates were definitely willing to consider TJA.However, patients' preferences for hip or knee replacements are strongly associated with their misperceptions of the indications for, and the risks and benefits of, these procedures. These misperceptions can be corrected with the use of patient decision aids. Therefore, patient decision aids may have a role in ensuring that wait list reforms address under-use of surgical procedures that informed patients need and want, while preventing the over-use of procedures that informed patients do not value. If they were used in combination with screening for surgical eligibility, they might also prevent inappropriate referrals for surgery (i.e., patients who are not clinically eligible or who would not want surgery even if they were clinically eligible).

Objective:

To pilot test the feasibility of a trial evaluating the incremental effects of patient decision aids on reducing unnecessary surgical referrals for TJA, when used in combination with a general practitioner intake clinic that screens patients for surgical eligibility.

Participants & Setting:

Patients referred for surgical consultation for hip or knee osteoarthritis at The Ottawa Hospital will be recruited. Excluded are those with inflammatory arthritis, previous TJA, or those unable to understand video/DVD decision aids due to deafness, blindness, cognitive impairment, or language barrier.

Design:

In this pilot study, patients will be screened for surgical eligibility by a trained general practitioner using a standardized examination of the hip/knee and questionnaire assessing joint symptoms and disability. Eligible patients will be stratified by affected joint (hip/knee) and randomly allocated to either: a) usual education; or b) a patient decision aid which presents balanced evidence-based information on the treatment options, including the risks and benefits. Automated reports will be sent to the surgeon for all patients.

Primary Outcomes:

* Feasibility of participant recruitment, intervention provision, and data collection; sample size needed to detect differences in the rates of unnecessary referral

Secondary Outcomes

* Wait times to decision
* Knowledge
* Decision quality, the extent to which patients' decisions are informed and values-based.
* Decisional conflict

Timeline and Deliverables:

By the end of this one year study, we will prepare a report and policy brief on the evidence of feasibility to support a larger scale multi-centre trial and a fully implementable set of interventions, with standardized training, to facilitate replication elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for surgical consultation for hip or knee osteoarthritis at The Ottawa Hospital will be recruited

Exclusion Criteria:

* Patients with inflammatory arthritis
* Previous TJA
* Those unable to understand video/DVD decision aids due to deafness, blindness, cognitive impairment, or language barrier.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Stacey, PHD, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stacey D, Hawker G, Dervin G, Tomek I, Cochran N, Tugwell P, O'Connor AM. Management of Chronic Pain: Improving shared decision making in osteoarthritis. BMJ. 2008 Apr 26;336(7650):954-5. doi: 10.1136/bmj.39520.701748.94. Epub 2008 Apr 8. PMID 18397937
- [Result] Stacey D, Hawker G, Dervin G, Tugwell P, Boland L, Pomey MP, O'Connor AM, Taljaard M. Decision aid for patients considering total knee arthroplasty with preference report for surgeons: a pilot randomized controlled trial. BMC Musculoskelet Disord. 2014 Feb 24;15:54. doi: 10.1186/1471-2474-15-54. PMID 24564877
- See also: Clinical and Decision Summary tool — http://www.bmj.com/cgi/content/full/336/7650/954-a?view=long&pmid=18397937

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Patient Decision Aid: Patient decision aid about treatment options for osteoarthritis
  1. Patient decision aid: Patients will receive:
     i)patient education booklet ii) a video/DVD PtDA for either hip (Treatment choices for hip osteoarthritis) or knee (Treatment choices for knee osteoarthritis) © Health Dialog 2005.
     iii) a personal decision form is an interactive form used by patients after the DVD to elicit their knowledge, values, preferred option, and perceptions of the decision making process.
     iv) Referral to the surgeon with a standardized report of their clinical findings plus decisional data (knowledge, values, preference).
  2. Usual care: Patient will be given i) education booklet from local hospital which is a standardized teaching booklet given to all patients describing preparation for surgery, recovery after surgery, discharge plans.
  ii) Referral to the surgeon with a standardized report of their clinical findings.
- 2 Usual Care: Usual patient educational materials
  2 Usual care: Patient will be given i) education booklet from local hospital which is a standardized teaching booklet given to all patients describing preparation for surgery, recovery after surgery, discharge plans.
  ii) Referral to the surgeon with a standardized report of their clinical findings.
Period: Overall Study
Arm/Group | 1 Patient Decision Aid | 2 Usual Care
Started | 71 | 71
Completed | 69 | 71
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Patient Decision Aid | 2 Usual Care | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There was missing data for 3 patients in the usual education (control) arm of the study and missing data for 2 patients in the patient decision aid arm who dropped out of the study
  years
    number analyzed (Participants) | 69 | 68 | 137
    (all) | 67.1 (10.85) | 67.3 (12.16) | 67.2 (11.51)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: There was missing data for 2 patients in the patient decision aid arm who dropped out of the study
  Participants
    Gender: number analyzed (Participants) | 69 | 71 | 140
    Gender: Men | 19 | 25 | 44
    Gender: Women | 50 | 46 | 96
Region of Enrollment [Number; unit: participants]
  Canada | 71 | 71 | 142
Education Achieved [Count of Participants; unit: Participants] — Population: missing data - patients did not respond to the question on the survey or dropped out of the study
  Participants
    Less than secondary school | 10 | 12 | 22
    Secondary school/trades school | 25 | 30 | 55
    post-secondary education (e.g., university) | 32 | 24 | 56
    missing | 4 | 5 | 9
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) [Mean (Standard Deviation); unit: units on a scale] — A disease specific tool used for people with hip or knee osteoarthritis to measure physical function, pain and stiffness in the last 48 hours. It is self-administered with 24 items. Higher points signify higher levels of functional difficulty. The scores are summed for items with total score range of 0 to 96. For subscales, the possible ranges are as follows: pain=0-20, stiffness=0-8, physical function=0-68. Population: There was missing data for 2 patients in the patient decision aid intervention arm and 3 patients in the usual education arm.
  units on a scale
    number analyzed (Participants) | 69 | 68 | 137
    (all) | 60 (0.17) | 64 (0.18) | 62 (0.176)
Hip-Knee Priority Tool (HKPT) [Mean (Standard Deviation); unit: units on a scale] — Clinician assess patients for: pain on motion (none [0 points], mild [0], moderate [6], severe [13]), pain at rest (none [0], mild [3], moderate [8], severe [11]), ability to walk (>5 blocks [0], 1-5 blocks [0], <1 block [4], household ambulatory [7]), other functional limitations (none [0], mild [4], moderate [11], severe [19]), threat to independence (none [0], not immediate [10], immediate [20]), abnormal physical examination (none [0], mild [0], moderate [5], severe [10]), radiographic evidence (normal [0], abnormal [check]). Score is 0 (no limitations) to 80 (severe limitations). Population: There was missing data for 2 patients in the patient decision aid arm who dropped out of the study and for 3 patients in the usual education
  units on a scale
    number analyzed (Participants) | 69 | 68 | 137
    (all) | 43.9 (12.4) | 45.1 (17.5) | 44.5 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Data Collection at Month 12
Description: Feasibility was the number of participants who completed data collection at 12 months
Time Frame: Data collection occurred at month 12
Population: Two in the intervention group withdrew from the study and 3 in the control group were lost to follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Patient Decision Aid Intervention: Participants were given the patient decision aid plus usual education materials
- Usual Education (Control): Participants were only given usual education materials
Arm/Group | Patient Decision Aid Intervention | Usual Education (Control)
Number analyzed (Participants) | 69 | 68
Participants
  Surgery | 55 | 48
  Non-surgery management | 5 | 9
  Waiting list for surgery | 8 | 10
  Died | 1 | 1

2. Secondary Outcome: Wait Times
Description: length of time from screening consultation to a definitive decision - underwent surgery or off the wait list for non-surgical management
Time Frame: Data collection occurred at surgeon consult and month 12.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Patient Decision Aid Intervention | Usual Education (Control)
Number analyzed (Participants) | 69 | 71
weeks | 33.4 [26.0 to 41.4] | 33.0 [26.1 to 39.9]

3. Secondary Outcome: Participant's Knowledge
Description: The participants' knowledge was measured using 4-multiple choice questions (e.g., osteoarthritis progress over time, need for revision joint replacement, proportion of patients with reduced pain, length of time for recovery) taken from the Hip-Knee Osteoarthritis Decision Quality Instrument. The total score range was 0 to 4 based on correct responses to the questions. Higher score was higher knowledge.
Time Frame: Data collection occurred at week 2
Population: participants who completed the knowledge test after receiving the intervention/control intervention
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Patient Decision Aid Intervention | Usual Education (Control)
Number analyzed (Participants) | 66 | 66
percentage of correct answers | 71.2 (23.7) | 46.6 (21.4)

4. Secondary Outcome: Number of Participants With Sufficient Decision Quality
Description: Decision quality was deemed sufficient if a patient scored 66% or higher on the knowledge test (measured at 2 weeks) and if their predicted probability of surgery based on values corresponded with their actual choice (measured at 12 months). Values measured were from the Hip-Knee Osteoarthritis Decision Quality Instrument (measured at 2 weeks). Patients' values were measured by asking patients to rate the personal importance of the benefits and harms of outcomes for 6 items (e.g., relief of pain) on a 10 point rating scale with 1 indicating low importance and 10 indicating high importance. The match between the patients' choice and their values for benefits/risks was calculated as a dichotomous measure. The predicted probability of surgery was calculated for each patient using a logistic regression equation derived from three items assessing the patient's values. The equation was [1 + exp (-S)]-1 where S = -0.338
Time Frame: Data collection occurred at week 2 (knowledge and values) and month 12 (patients' chosen option).
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Decision Aid Intervention | Usual Education (Control)
Number analyzed (Participants) | 55 | 56
Participants | 31 | 14

5. Secondary Outcome: Number of Participants With no Decisional Conflict
Description: SURE test version of the Decisional Conflict Scale was used to measure no decisional conflict. This scale is called the SURE test and has 4 items. Total score range is 0 to 4 and a score of 4 indicates no decisional conflict. Any score less than 4 indicates decisional conflict.
Time Frame: Data collection occurred at week 2
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Decision Aid Intervention | Usual Education (Control)
Number analyzed (Participants) | 65 | 66
Participants | 45 | 38

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patient Decision Aid Intervention | Usual Education (Control)
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/71
Other Adverse Events (participants affected / at risk) | 0/69 | 0/71

LIMITATIONS AND CAVEATS:
Patients need to be followed for longer given that 13% were still waiting for surgery after one year.

Decisional conflict and preferred option were only measured prior to seeing the surgeon.

Limitations related to the preliminary effectiveness outcomes are potential for self-report bias given that most outcome measures were patient reported. For actual choice, self-report bias may have been mitigated because data was also extracted from the patients' health record for verification of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No